CLINICAL TRIAL: NCT07394296
Title: Study of the Prevalence of Midline Replacements and the Reasons for These Replacements
Acronym: MIDRELAY
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Other Study IDs: 2025-03-01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Veinous Access; Midline; Veinous Capital
Keywords: midline; midline placement; midline indication; patient care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 33 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Venous access management plays a key role in patient care and preserving their venous capital. The so-called "conventional" peripheral venous catheter is the most common venous access device, but it is associated with a high rate of complications, particularly in cases of prolonged use or poor venous capital. Recommendations, such as those from MAGIC or SF2H, advocate their use when the intended duration of use is 5 days or less. For longer periods or in cases of difficult access, so-called "central" devices such as PICC lines or central venous catheters are used, although they present specific risks such as CLASBI or deep vein thrombosis.

In intermediate situations, the midline, a peripheral venous access device, is a relevant alternative, particularly for non-venotoxic intravenous treatments lasting more than 5 days. Although it is theoretically associated with fewer infections and complications than the PICCline, its complication rate and actual duration of use vary widely in the literature.

The MAGIC recommendations suggest using them for periods of 14 days or less. The widespread use of midlines in healthcare facilities, and in particular the creation of vascular access units, has given rise to issues shared between centers, notably the replacement rate of these devices. The study therefore aims to determine the replacement and early removal rates for midlines, the circumstances in which they are replaced, and toassess the relevance of the 28-day limit in the choice of device, in order to improve practices and optimize the practitioner's initial decision.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients who have given their consent to participate in the study.
* Patients treated in a hospital unit authorized to insert midlines, or who have a midline inserted by a professional trained in this procedure, in accordance with the local organization of each center.
* First insertion for the treatment of a given event with an expected treatment duration of 28 days or less.
* Patients treated with a midline catheter at least 14 cm in length.

Exclusion Criteria:

* No coverage by the social security system
* Failure to insert the midline
* Patient under guardianship or conservatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study are those whose midline indication has been validated by the vascular access unit according to the hospital's organization. The expected duration of midline use should be 28 days or less.
Sampling Method: Probability Sample
Enrollment: 984 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the midline replacement rate regardless of the indication, in the various requesting centers | within 28 days after the initial placement of the midline
  The primary endpoint is the cumulative incidence rate of midline replacement over a censored period of 28 days. This period begins on the day of inclusion with the first midline placement, regardless of the indication. Competing events are removal without replacement, regardless of the cause (death, removal at the end of treatment, early removal before the end of treatment without replacement).

SECONDARY OUTCOMES:
Secondary objective 1: To evaluate the early removal rate among patients living with midlines within 28 days of placement. | over a censored period of 28 days
  Cumulative incidence rate of early removal of midlines placed on the day of inclusion over a censored period of 28 days. Competing events are death and removal due to end of treatment
Secondary objective 2: Describe the reasons for early removal of midlines. | Withdrawals are analyzed from the day of inclusion and over a censored period of 28 days
  Midline removal rate for each of the following reasons:
  * Extravasation/diffusion of the product
  * Suspected midline infection
  * Confirmed midline infection
  * Accidental removal
  * Catheter-induced deep vein thrombosis
  * Catheter occlusion
  * Inability to perform sampling
  * Conversion to PICCline
  * Duration exceeded
Secondary objective 3: Describe the lifespan of midlines | This duration includes the number of days between the day of inclusion and the day of device removal over a censored period of 28 days.
  Midline lifespan. The event is the removal of the midline regardless of the cause: removal at the end of treatment, removal due to death, early removal (with or without reinsertion).
Secondary objective 4: Describe the replacement rate of midlines among midlines still in place at different time | Days 7, 14, 21 and 28
  Cumulative incidence rate of midline recurrence with a benchmark at D7, D14, then D21, censored at D28
Secondary objective 5: Compare the midline replacement rate between the initial indication of antibiotic therapy and the initial indication of insufficient venous capacity | Replacements taken into account occur over a censored period of 28 days beginning on the day of inclusion
  Cumulative incidence rate of midline removal for the initial indication of antibiotic therapy and midline removal rate for the initial indication of insufficient venous access. The midlines analyzed are those placed on the day of inclusion. Concurrent events are removal without replacement regardless of the cause (death, removal at the end of treatment, early removal before the end of treatment without replacement).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, France